CLINICAL TRIAL: NCT03290872
Title: A Study to Assess the Effects of Two Commonly Used Mitral Valve Annuloplasty Rings in Mitral Valve Repair on Short-term Outcomes.
Brief Title: Mitral Annuloplasty Rings RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-7851
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Degenerative Mitral Valve Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carpentier Edwards Physio 2 Complete flexible mitral ring (Active Comparator): Mitral Valve Annuloplasty Ring Repair using Carpentier Edwards Physio 2 Complete flexible mitral ring
  Interventions: Device: Carpentier Edwards Physio 2 Complete flexible mitral ring
- Simplici T Partial flexible mitral annuloplasty ring (Active Comparator): Mitral Valve Annuloplasty Ring Repair using Simplici T Partial flexible mitral annuloplasty ring
  Interventions: Device: Simplici T Partial flexible mitral annuloplasty ring

INTERVENTIONS:
Device: Carpentier Edwards Physio 2 Complete flexible mitral ring — Mitral valve Annuloplasty Ring repair using a Carpentier Edwards Physio 2 Complete flexible mitral ring
  Arms: Carpentier Edwards Physio 2 Complete flexible mitral ring
Device: Simplici T Partial flexible mitral annuloplasty ring — Mitral valve Annuloplasty Ring repair using a Simplici T Partial flexible mitral annuloplasty ring
  Arms: Simplici T Partial flexible mitral annuloplasty ring

SUMMARY:
Recently published work has suggested that mitral valve annuloplasty ring type may affect the development of post-repair mitral stenosis resulting in adverse intracardiac hemodynamics and poor functional status. However, these results have not been comprehensively determined in a systematic manner on a general mitral valve repair population. As well, an underlying mechanism for these findings is not understood.

The investigators hypothesize that mitral valve repair with a complete annuloplasty ring (Carpentier-Edwards Physio II) when compared to repair with a partial annuloplasty ring (Simplici- T) may not necessarily result in elevated mitral gradients consistent with functional mitral stenosis (FMS). Currently no prospective data exists to test the hypothesis that a correctly sized, flexible complete annuloplasty ring has detrimental effects.

As 60% of annuloplasty rings used in surgical repair of degenerative mitral valve disease in North America utilizes one of the many forms of complete flexible rings available, this information is urgently required.

The investigators will evaluate: 1) the effect on mitral valve hemodynamics, 2) changes to mitral annular, valvular and subvalvular structure and function with 3D echocardiography, and 3) the effect on patient functional capacity at 1 year.

If FMS early post repair is a real phenomenon, the investigators hope to better understand the mechanisms through the use of advanced imaging techniques-namely 3D modeling of the mitral valvular apparatus, aortic mitral interactions and LV remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Mitral regurgitation secondary to degenerative valve disease referred to Prof Tirone David (Co-investigator) will be invited to take part.
* The mitral valve anatomy must be anatomy suitable for repair.
* The patient must be able to perform treadmill exercise echocardiography.
* The patient must be over 18 years of age.

Exclusion Criteria:

* Any presence of life-limiting disease process, for example advanced malignancy.
* Hemodynamically unstable patients in cardiogenic shock
* Concomitant aortic valve disease/surgery
* Previous mitral valve repair
* Impaired left ventricular systolic function as defined by a left ventricular ejection fraction of ≤ 50%.
* If the patient lives out of state or cannot attend follow up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Mean mitral valve gradient | 1 year
  Mean mitral valve gradient measured by transthoracic echocardiogram

SECONDARY OUTCOMES:
Left ventricular remodelling | 1 year
  Assessment of left ventricular remodelling obtained from transthoracic echocardiography performed pre-operatively and at 1 year post surgery using 3D LV end-diastolic volume and 3D end-systolic volume measurements and 3D LV ejection fraction
Aortic-mitral coupling | 1 year
  3D transesophageal echocardiogram assessment intra-operatively both pre and post bypass assessing the entire mitral valvular and subvalvular apparatus, the left ventricle and the aortic valve to assess aortic-mitral valvular coupling and to determine whether there is a difference observed in aorto-mitral coupling between complete and partial ring repairs
Change in functional capacity | 1 year
  Functional capacity will be specifically assessed using workload achieved on stress transthoracic echocardiogram studies performed pre surgery and at 1 year post surgery. Measurements acquired will include total exercise time and total workload achieved. Also patients will complete SF-36 questionnaires pre-surgery and at 1 year post surgery for further assessment of change in functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Wendy W Tsang, MD, Principal Investigator — University Health Network, Toronto General Hospital

IPD SHARING:
Plan to Share IPD: No